CLINICAL TRIAL: NCT00761488
Title: Recommendations for Monitoring Clinical Experience Following Implantation of the AcrySof® Toric
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Primary Investigator resigned from hospital
Sponsor: Alcon Research (Industry)
Responsible Party: Ricky Ho, RA Manager, Alcon Research Ltd.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HK-Toric-YIU-01
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2010-01

CONDITIONS: Cataract
Keywords: Visual acuity,; corneal and; refractive; cylinder; following; implantation of the; AcrySof® Toric
MeSH Terms: conditions — Cataract

ARMS (1):
- 1 (Experimental): AcrySof® Toric IOL
  Interventions: Device: AcrySof® Toric IOL

INTERVENTIONS:
Device: AcrySof® Toric IOL — Implanted into the study eye

SUMMARY:
To allow surgeons to obtain clinical experience on the postoperative uncorrected and best distance corrected visual acuities (UCVA and BDCVA) and corneal and refractive cylinder of the AcrySof Toric IOL.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years old; of any race and gender; diagnosed with bilateral cataracts; require cataract extraction followed by implantation of a posterior chamber IOL; patients have between 0.75 -2.5 D of astigmatism preoperatively as measured by K readings.

Exclusion Criteria:

* Females of child bearing potential;irregular corneal astigmatism;keratopathy/Keratectasia; cornea inflammation or edema;previous corneal reshaping,dystrophy or transplant;amblyopia;glaucoma;RPE/Macular changes;diabetic retinopathy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Corneal astigmatism; IOL rotation | Before opertation; 1 day following implantation of each eye; 1, 3 months following lens implantation in the second eye.

SECONDARY OUTCOMES:
Uncorrected and best distance corrected visual acuities (UCVA and BDCVA) | Before opertation; 1 day following implantation of each eye; 1, 3 months following lens implantation in the second eye.

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States